CLINICAL TRIAL: NCT04890366
Title: Combination of the Immune Modulator Dimethyl Fumarate With Alteplase in Acute Ischemic Stroke
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: haojunwei3
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Dimethyl Fumarate; immune modulator; Alteplase; Acute Ischemic Stroke; edema
MeSH Terms: conditions — Ischemic Stroke; Edema | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alteplase plus Dimethyl Fumarate (Experimental)
  Interventions: Drug: Dimethyl Fumarate
- Alteplase (No Intervention)

INTERVENTIONS:
Drug: Dimethyl Fumarate — Dimethyl fumarate 240mg orally twice daily for 3 consecutive days
  Arms: Alteplase plus Dimethyl Fumarate

SUMMARY:
The investigators conduct this study to investigate whether oral administration of Dimethyl Fumarate, a Food and Drug Administration-approved drug for multiple sclerosis, is safe and effective in combination with alteplase in patients with Acute Ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

1. more than 18years old
2. NIHSS score≥5
3. MRI shows anterior circulation infarction
4. Patients who meet Alteplase thrombolytic therapy within 4.5h
5. The time from onset to DMF application was less than 24 hours

Exclusion Criteria:

1. Hemorrhagic stroke
2. Patients who have received or plan to receive endovascular therapy
3. Other diseases of the central nervous system
4. Pre-existing neurological disability (mRS Score >2)
5. Vertebrobasilar artery obstruction
6. Difficulty swallowing
7. Patients who cannot accept MRI examination
8. Abnormal liver function (transaminase higher than 2 times the normal upper limit)
9. The lymphocyte count was lower than the lower limit of normal value
10. Anti-tumor drugs, other immunosuppressive and immunomodulatory drugs are being used
11. Patients known to have hypersensitivity to dimethyl fumarate or any excipients
12. Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in lesion volume | baseline to day 7
  measured by MRI
changes in hemorrhage volume | baseline to day 7
  measured by MRI
changes in National Institutes of Health Stroke Scale (NIHSS) | baseline to day 7
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.

SECONDARY OUTCOMES:
The Modified Rankin Scale (mRS) | day1
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day3
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day7
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day14
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day90
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
National Institutes of Health Stroke Scale (NIHSS) | day 3
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 7
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 14
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day 90
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, PhD,MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China